CLINICAL TRIAL: NCT01571986
Title: Improving Non Invasive Ventilation
Brief Title: Improving Non-invasive Ventilation
Acronym: Improving NIV
Status: Recruiting | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, Principal Investigator, Università Vita-Salute San Raffaele
Other Study IDs: VP/50/ER/mm
Record Dates: First submitted 2012-03-16; First posted 2012-04-05 (Estimated); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Acute Respiratory Failure
Keywords: NIV; acute respiratory failure; hypoxia; hypercapnia; non-invasive ventilation; hospital ward
MeSH Terms: conditions — Hypoxia; Hypercapnia | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NIV: All patients with acute respiratory failure treated with non-invasive ventilation who give informed consent about treatment of their clinical data
  Interventions: Procedure: Non-invasive ventilation

INTERVENTIONS:
Procedure: Non-invasive ventilation — Non-invasive ventilation

SUMMARY:
A single center, observational, prospective study to improve knowledge about non-invasive ventilation, obtaining data about compliance, efficacy, imaging in patients who already receive non-invasive ventilation as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* treatment with non-invasive ventilation
* informed consent

Exclusion Criteria:

* refusal of informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with acute respiratory failure treated with non-invasive ventilation who give informed consent about treatment of their clinical data
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients requiring NIV in a large university hospital. Incidence of NIV failure (including patient compliance) and NIV related complications. Imaging (chest ultrasound) in a subgroup of patients before and after receiving NIV. | Outcome measures will be assessed every day and participants will be followed for the duration of hospital stay, an expected average of 1 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele di Milano, Milan, Italy

REFERENCES:
- [Background] Cabrini L, Nobile L, Plumari VP, Landoni G, Borghi G, Mucchetti M, Zangrillo A. Intraoperative prophylactic and therapeutic non-invasive ventilation: a systematic review. Br J Anaesth. 2014 Apr;112(4):638-47. doi: 10.1093/bja/aet465. Epub 2014 Jan 19. PMID 24444661
- [Background] Cabrini L, Plumari VP, Nobile L, Olper L, Pasin L, Bocchino S, Landoni G, Beretta L, Zangrillo A. Non-invasive ventilation in cardiac surgery: a concise review. Heart Lung Vessel. 2013;5(3):137-41. PMID 24364004